CLINICAL TRIAL: NCT05799352
Title: Effects of Endoscopic Lung Volume Reduction on Diaphragm Function and Conformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Olivier Taton, Doctor, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2018/227
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Intervention Model Description: Before and after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endoscopic lung volume reduction (Experimental): All the patients will have endobronchial valves insertion. We will evaluate before and 3 months after the evolution of the diaphragmatic strength and conformation.
  Interventions: Device: Endoscopic lung volume reduction

INTERVENTIONS:
Device: Endoscopic lung volume reduction — a prospective monocentric study on hyperinflated COPD patients without collateral ventilation. Patients were evaluated before and 3 months after unilateral ELVR by transdiaphragmatic pressure (Pdi) measured at the functional residual capacity (FRC) after magnetic phrenic stimulation and by high-resolution computed tomography at the FRC allowing 3D modelling of the diaphragm for measurements of fibers length, length of the zone of apposition and radius of curvature of the diaphragmatic domes.

SUMMARY:
Chronic obstructive lung disease (COPD) is a common disease that is frequently complicated by hyperinflation. The resulting increase in lung volume impairs the diaphragmatic function because of a shortening of the diaphragmatic fibers and an increase in the radius of curvature of the diaphragmatic domes. Lung volume reduction surgery (LVRS) has already shown an improvement in diaphragmatic function that could be explained by a change of the diaphragm conformation. More recently, endoscopic lung volume reduction (ELVR) has shown benefits in terms of respiratory function, exercise capacity and quality of life, but the mechanisms of these improvements are poorly understood. Therefore, we aim to evaluate the evolution of the diaphragmatic function and the changes in diaphragmatic conformation after unilateral ELVR.

ELIGIBILITY:
Inclusion Criteria:

* valves insertion

Exclusion Criteria:

* TLVR < 50 %

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Transdiaphragmatic pressure | before until 3 months after the valves insertion
  evaluate the difference in diaphragmatic function, assessed by the transdiaphragmatic pressure, before and 3 months after unilateral valves setting
Diaphragmatic conformation | before until 3 months after the valves insertion
  evaluate the change of the diaphragm conformation, by measuring diaphragmatic fibers length in several planes, diaphragmatic area and radius of curvature, before and 3 months after unilateral ELVR.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Taton, Principal Investigator — Hôpital Erasme, Université Libre de Brussels, Brussels, Belgium
Locations (1):
- Erasme Hospital, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taton O, Perez-Bogerd S, Van Muylem A, Gevenois PA, Van Hove O, Bondue B, Brenard E, Leduc D. Chest mechanics after endoscopic lung volume reduction: Comparison between responders and non-responders based on dynamic hyperinflation. Respir Med Res. 2025 Nov;88:101194. doi: 10.1016/j.resmer.2025.101194. Epub 2025 Jul 23. PMID 40763652
- [Derived] Taton O, Gevenois PA, Van Muylem A, Bondue B, Van Laethem S, Leduc D. Improvements of the shape and strength of the diaphragm after endoscopic lung volume reduction. Thorax. 2024 Jul 16;79(8):711-717. doi: 10.1136/thorax-2024-221375. PMID 38914469